CLINICAL TRIAL: NCT03887559
Title: Adding a Group Based Stabilization and Skill Training Intervention for Patients With Long Lasting Posttraumatic Reactions Receiving Outpatient Treatment in Specialized Mental Health Care - A Randomized Controlled Trial
Brief Title: Group-based Stabilization and Skill Training for Patients With Lasting Posttraumatic Reactions in Mental Health Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/957
Record Dates: First submitted 2019-03-11; First posted 2019-03-25 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Stress Disorders, Post-Traumatic; Mental Disorders; Trauma and Stressor Related Disorders
Keywords: Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Mental Disorders; Trauma and Stressor Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Group-based stabilization and skill-training combined with individual treatment.
  Interventions: Behavioral: Group-based stabilization and skill training in addition to individual treatment
- controls (Active Comparator): Individual treatment as usual only.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Group-based stabilization and skill training in addition to individual treatment — Group-based stabilization and skill training, weekly 2-hour sessions during 20 weeks. Based on the manual "Tilbake til Nåtid" ("Back to here and now") (Holbæk, 2014) developed by clinicians in the highly specialized national trauma clinic 'Modum Bad's Trauma Clinic'.
  Arms: Intervention group
Other: Treatment as usual — Treatment as usual: conventional individual treatment (outpatient). Not standardized.
  Arms: controls

SUMMARY:
This study evaluates the addition of a group based stabilization and skill-training intervention to individual out-patient treatment for long lasting post-traumatic reactions. Half of the participants will receive the combined treatment while the other half will receive individual treatment as usual.

DETAILED DESCRIPTION:
Many patients in mental health care have previously experienced life-stressors and traumatic events that are related to the problems they seek treatment for. Although the diagnostic labels vary, the clinical picture often demonstrates long lasting complex psychological and somatic post-traumatic symptoms such as avoidance, bodily activation, difficulties in regulating emotions and in relationships with others, impaired quality of life and reduced level of function. Patients often receive long-term individual therapy in general mental health care, occasionally without clinically significant improvement. Still, they continue treatment due to high symptom pressure and low level of functioning. The study targets a novel intervention which tests the effect of adding a group based stabilization and skill training intervention to conventional individual treatment among 160 patients already receiving treatment in a community mental health hospital. Change in variables covering mental health issues, functional impairment, well-being, use of hospital services and drug prescriptions will be examined, as well as markers of inflammation found in sera before and after intervention. The purpose is to develop better and more effective treatment options for a large number of patients who receive mental health care in community mental health hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment in ordinary out-patient clinics
* Having been exposed to or witnessing to traumatic event(s) defined as "one or several extremely threatening or horrific events or series of events or situations being of such a character which is likely to overwhelming distress in almost anyone in a similar situation", measured by Stressful Life Events Screening Questionnaire
* Presenting with posttraumatic reactions such as hyperarousal, avoidance, intrusions, emotional dysregulation or interpersonal difficulties.
* Symptom duration for a minimum of six months.
* Understand and speak Norwegian to an extent that is required to participate in a stabilization- and skill-training group.

Exclusion Criteria:

* Active psychotic symptoms.
* Substance or drug addiction or abuse.
* High suicidal risk considered by the individual therapist.
* Having participated in the course previously.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Questionnaire about Process of Recovery' (QPR) Change from baseline | 4 weeks after intervention group has completed group treatment
  Experienced personal recovery is measured by self-report; 'Questionnaire about Process of Recovery' (QPR)
Questionnaire about Process of Recovery' (QPR) Change from baseline | 6 months after intervention group has completed group treatment
  Experienced personal recovery is measured by self-report; 'Questionnaire about Process of Recovery' (QPR)
Questionnaire about Process of Recovery' (QPR) Change from baseline | 12 months after intervention group has completed group treatment
  Experienced personal recovery is measured by self-report; 'Questionnaire about Process of Recovery' (QPR)

SECONDARY OUTCOMES:
The Work and Social Adjustment Scale (WSAS) change from baseline | 4 weeks, 6 months and 12 months after intervention group has completed group treatment
  Functional impairment associated with mental Health measured by self-report
The International Trauma Questionnaire (ITQ) change from baseline | 4 weeks, 6 months and 12 months after intervention group has completed group treatment
  Self-report to capture elements of post-traumatic stress disorder (PTSD) and complex post-traumatic stress disorder (CPTSD)
The Clinical Outcome in Routine Evaluation (CORE-10) change from baseline | 4 weeks, 6 months and 12 months after intervention group has completed group treatment
  Sel-report measure of psychological distress, capturing general mental health issues.
WHO Five Well-Being Index (WHO-5) change from baseline | 4 weeks, 6 months and 12 months after intervention group has completed group treatment
  Questionnaire assessing subjective psychological well-being and also a measure of depression.
Posttraumatic Cognition Inventory (PTCI-9) change from baseline | 4 weeks, 6 months and 12 months after intervention group has completed group treatment
  Self-report measure of negative and dysfunctional posttraumatic cognitions

OTHER OUTCOMES:
Use of health services in hospitals - Data extracted from The National Patient Register (NPR)- change from baseline | 12 months after group intervention
  The National Patient Register (NPR) regularly receives data from all health authorities in Norway on treatment episodes in hospitals and mental health services. Data extracted will include type of clinical unit, time of admission, length of stay in inpatient units, consultations in outpatient units and mobile teams and diagnoses, measured 12 months before group intervention and 12 months after group intervention.
Prescriptions of medicine -Data extracted from The Norwegian Prescription Database - change from baseline | 12 months after group intervention
  The Norwegian Prescription Database regularly receives data on prescriptions on drug prescriptions from doctors in primary and secondary health care services and hospitals. Extracted data will cover prescriptions, 12 months before group intervention and 12 months after group intervention.
Occupational status- Data extracted from The Norwegian Labour and Welfare Administration (NAV)- change from baseline | 12 months after group intervention
  The Norwegian Labour and Welfare Administration (NAV) have data on all citizens working status and sick-leaves lasting for more than two weeks. Extracted data will include information such as sick- and disability leaves 12 months before group intervention and 12 months after group intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Lise Løvaas, Study Director — St. Olavs Hospital
Locations (1):
- Department of Tiller DPS, St. Olavs Hospital University Hospital in Trondheim, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holgersen KH, Bronstad I, Jensen M, Brattland H, Reitan SK, Hassel AM, Arentz M, Lara-Cabrera M, Skjervold AE. A combined individual and group-based stabilization and skill training intervention versus treatment as usual for patients with long lasting posttraumatic reactions receiving outpatient treatment in specialized mental health care - a study protocol for a randomized controlled trial. Trials. 2020 May 27;21(1):432. doi: 10.1186/s13063-020-04297-z. PMID 32460840